CLINICAL TRIAL: NCT04756258
Title: Early Diagnosis of Leukemic Children Patients Based on Clinical, Age Estimation and Radiographical Evaluation of Oral Affection
Status: Completed | Type: Observational
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, rehab ghouraba, lecturer, Tanta University
Other Study IDs: 222
Record Dates: First submitted 2021-02-08; First posted 2021-02-16 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Leukemia
MeSH Terms: conditions — Leukemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Early diagnosis of leukemia which is malignant tumor affecting bone especially in children is import to allow early intervention improving prognosis. It is known that leukemic patients suffer from clinical signs as anemia, thrombocytopenia, and pronounced hepatosplenomegaly or lymphadenopathy. However, sometimes these clinical signs may be not clearly manifested and may look like anemia. The early diagnosis could be achieved through dentist by accessing clinical and radiographical signs such as oral masses, gingival bleeding /or enlargement and oral ulceration with radiographical features including focal or generalized osteolysis of bone with presence of moth eating appearance and even with abnormal teeth chronology regarding teeth morphology, germ formation of permanent teeth and their sequence of eruption. Therefore, accessing of these special clinical and radiographical features by the dentist could help in early diagnosis of leukemic children patients

DETAILED DESCRIPTION:
Ten children patients suffer from leukemia selected after initial diagnosis from hematology unit of faculty of medicine, Tanta university based on their clinical signs such as; bone pain, fatigability, lymph node enlargement…etc., with abnormal CBC revealing anemia or abnormal WBCs. These patients accessed clinically for oral signs and accessed radiographically using panoramic radiographs and cone beam computed tomography (CBCT) to evaluate chronology and bone density.

ELIGIBILITY:
Inclusion Criteria:

1-Children will be aged from 6-10 years 2 Children diagnosed with leukemia but they don't start treatment yet

-

Exclusion Criteria:

1. Children below or above the age
2. Children already diagnosed by leukemia and started treatment
3. Children diagnosed by other bone lesions showing osteolytic bone or anemia as thalassemia or sickle cell anemia or any other bone pathology

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: ten Children leukemic patients selected from hematology Unit of faculty of medicine, Tanta university revealing anemia or abnormal WBCs confirmed by bone marrow aspiration biopsy, these Children patients examined orally for any oral pathology as gingival masses, oral ulceration, bone resorption, teeth mobility, and assessed radiographically by panoramic and CBCT for age estimation , bone density to help in their early diagnose if they came to the dentist
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2020-01-30 (Actual); Primary Completion 2020-10-22 (Actual); Study Completion 2020-10-22 (Actual)

PRIMARY OUTCOMES:
Ability to diagnose leukemic child patients who don't have manifesting systemic clinical signs from their clinical and radiographical oral signs | one year
  theses leukemic child patients could be diagnosed based on observation of oral signs such as oral masse, ulcers lake normal red hallow, bone loss around teeth without presence of local factors, abnormal teeth chronology regarding teeth morphology and eruption, germ formation of permanent teeth and their sequence of eruption and abnormal bone density through panoramic and CBCT images

CONTACTS AND LOCATIONS:
Overall Officials: rehab f ghouraba, PHD, Principal Investigator — Tanta university, faculty of dentistry, Oral medicine clinic; rehab f ghouraba, Principal Investigator — Tanta university, faculty of dentistry, Oral medicine clinic
Locations (1):
- Rehab Fouad Ghouraba, Tanta, Grabia, Egypt

IPD SHARING:
Plan to Share IPD: No